CLINICAL TRIAL: NCT03136107
Title: Determination of the Sun Protection Factor of a Cosmetic Daily Defence Skin Cream
Brief Title: Determination of the Sun Protection Factor (SPF) of a Cosmetic Daily De-fence Skin Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207640
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The trained grader responsible for assessing Minimal Erythemal Dose of unprotected skin (MEDu) and Minimal Erythemal Dose of product treated (MEDp) at Visit 5 will be blinded to the product allocation of subjects. The trained grader responsible for assessing the provisional MEDu at Visit 3 will, necessarily, not be blinded since only one test site will be exposed to Ultraviolet (UV) radiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test product (Experimental): This arm will include all the test sites on the participants back where test product (Physiogel Daily Defence Protective Day Cream Light) will be applied.
  Interventions: Other: Physiogel Daily Defence Protective Day Cream Light
- Reference product (Active Comparator): This arm will include all the test sites on the participants back where reference product (ISO 24444:2010 P3 standard sunscreen) will be applied.
  Interventions: Other: ISO 24444:2010 P3 Standard Sunscreen
- Negative control (No Intervention): This arm will include all the test sites on the participants back which will be left unprotected.

INTERVENTIONS:
Other: Physiogel Daily Defence Protective Day Cream Light — Investigator controlled, topical application to the epidermis at a dose of 2 milligrams per square centimeter (mg/cm2). Single application.
  Arms: Test product
Other: ISO 24444:2010 P3 Standard Sunscreen — Investigator controlled, topical application to the epidermis at a dose of 2 mg/cm2. Single application.
  Arms: Reference product

SUMMARY:
The purpose of this study is to determine the SPF of the test product according to the International Standards Organization (ISO) 24444:2010 methodology (In vivo determination of the SPF).

DETAILED DESCRIPTION:
A single-center, randomized, evaluator blind, intra-individual comparison, no treatment and positive controlled clinical study to determine the SPF of Physiogel Daily Defence Protective Day Cream Light as per ISO 24444:2010. The provisional minimal erythemal dose of unprotected skin (MEDu) for each subject will be determined before starting the test phase. Once the provisional MEDu for a subject has been determined, the three test sites will be demarcated. The test product and positive control (P3 reference sunscreen formulation) will be applied to two of the three test sites. The other test site will remain unprotected. All three test sites will be exposed to UV radiation at the expected MED and subsequently evaluated for erythema 16-24 hours after UV exposure.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination
* Subjects with a Fitzpatrick Skin Type of I, II or III
* Subjects with an Individual typological angle (ITA°) greater than 28°

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding or lactating
* Subjects having used medication with known photo-toxic and/or photosensitizing potential (e.g. hypericum perforatum, antibiotics, blood pressure regulating agents) up to 14 days prior to screening
* Subjects with a history of systemic therapy with anti-inflammatory agents or analgesics (e.g. diclofenac) up to 3 days prior to screening
* Subjects with dermatological conditions
* Subjects with a history of abnormal response to the sun
* Subjects who are tanned or have had sun exposure on the back area in the previous 4 weeks prior to screening
* Subjects having marks, blemishes or nevi or presenting existing sun damage in the test area
* Subjects having excessive hair, moles, tattoos, scars or other imperfections in the test area that could influence the investigation
* Subjects with a history of systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. anti-allergics) up to 7 days prior to screening
* Subjects with a non-uniform skin colour or hyperpigmentation in the test area
* Subjects with a medical history of dysplastic nevi or melanoma
* Subjects with one of the following illnesses that might require regular systemic medication: Insulin-dependent diabetes, cancer
* Subjects with asthma, unless medicated
* Subjects with an electronic implant (e.g. pace maker, insulin pump, hearing aid) that cannot be removed during irradiation
* Acquired immune deficiency syndrome (AIDS) and infectious hepatitis, if known to the subjects
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Known allergy to latex
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days prior to screening
* Participation in another clinical study involving UV exposure to the same test site up to 2 months prior to screening
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* Subjects who have used a tanning bed or other tanning treatment on the back area up to 1 month prior to screening
* Subjects accustomed to using tanning beds
* Subjects who have used self-tanning products on the back area in the previous 1 month prior to screening
* An employee of the sponsor or the study site or members of their immediate family
* Subjects who will turn 71 years old before completing all assessment visits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were randomized at one center in Germany.
Groups:
- All Participants: There were a total of 4 test sites assigned to each participant: 1) untreated skin for provisional MEDu assessment; 2) untreated skin for SPF assessment; 3) test product (Physiogel Daily Defence Protective Day Cream Light); and 4) reference product (ISO 24444:2010 P3 standard sunscreen). Test sites were delineated on the dorsum between the scapula and waist, either side of the spine. The test and reference products were applied topically to separate test sites by trained technician at a dose of 2 milligrams per square centimeter (mg/cm2) as per the randomization schedule. All participants who were randomized to receive the study treatments were included.
Period: Overall Study
Arm/Group | All Participants
Started | 26
Test Product | 26
Reference Product | 26
Negative Control | 26
Completed | 25
Not Completed | 1
Not completed — Other (Not specified) | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline population included safety population (N=26), safety population included all participants randomized and received any application of the study products.There were a total of 4 test sites assigned to each participant: 1) untreated skin for provisional MEDu assessment; 2) untreated skin for SPF assessment; 3) test product (Physiogel Daily Defence Protective Day Cream Light); and 4) reference product (ISO 24444:2010 P3 standard sunscreen). Test sites were delineated on the dorsum between the scapula and waist, either side of the spine. The test and reference products were applied topically to separate test sites by trained technician at a dose of 2 milligrams per square centimeter (mg/cm2) as per the randomization schedule.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Arithmetic Mean of Individual Sun Protection Factor (SPFi) Value
Description: Arithmetical mean of all valid SPFi values of each product on each participant was calculated from the individual Minimal Erythemal Dose (MED) on product treated (MEDp) test sites in relation to unprotected (MEDu) test sites 16-24 hours after exposure to ultraviolet (UV) radiation (SPFi = MEDp/MEDu). The Minimal Erythemal Dose (MED) was defined as the lowest dose of UV radiation that produced the first perceptible unambiguous erythema with defined borders appearing over most of the field of UV exposure, 16 to 24 hours after UV exposure. No inferential statistical analysis has been performed for this outcome. Test and reference products achieved a 95% CI of ±16.4% and ±16.6% of the mean SPF. These data meet the statistical criterion defined in ISO 24444:2010 as the 95% CI is within ±17% of the mean SPF.
Time Frame: Up to 24 hours post UV exposure
Population: Intent to treat (ITT, N= 25) all valid participants data with no major protocol deviations were included in the SPF calculations. All participants exposed to Ultra Violet (UV) radiation were included the safety population, irrelevant of whether they successfully complete the study.
Measure: Mean (95% Confidence Interval); unit: Ratio (unit less)
Groups:
- Test Product: This arm included all the test sites on the participants back where test product (Physiogel Daily Defence Protective Day Cream Light) was applied.
- Reference Product: This arm included all the test sites on the participants back where reference product (ISO 24444:2010 P3 standard sunscreen) was applied.
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 25 | 25
Ratio (unit less) | 19.4 [16.24 to 22.63] | 14.0 [11.70 to 16.36]
Statistical Analysis 1: Comparison: Test Product vs Reference Product; CI % values (which is the percentage that half the 95 % CI represents of the mean values); Test type: Equivalence — Statistical criterion defined in ISO 24444:2010 is that the 95 %CI is within ±17 % of the mean SPF; Test product CI of ±16.4% and reference product CI of ±16.6% of the mean SPF

ADVERSE EVENTS:
Time Frame: Approximately 17 days
Groups:
- Negative Control: This arm included all the test sites on the participants back which were left unprotected.
- All Participants: Safety population included all participants randomized and received any application of the study products.There were a total of 4 test sites assigned to each participant: 1) untreated skin for provisional MEDu assessment; 2) untreated skin for SPF assessment; 3) test product (Physiogel Daily Defence Protective Day Cream Light); and 4) reference product (ISO 24444:2010 P3 standard sunscreen). Test sites were delineated on the dorsum between the scapula and waist, either side of the spine. The test and reference products were applied topically to separate test sites by trained technician at a dose of 2 milligrams per square centimeter (mg/cm2) as per the randomization schedule.
Arm/Group | Test Product | Reference Product | Negative Control | All Participants
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03136107/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03136107/SAP_001.pdf